CLINICAL TRIAL: NCT04196868
Title: Randomized Placebo-controlled Trial Comparing Methotrexate vs. Methotrexate/Metformin Association in Rheumatoid Arthritis Patients
Brief Title: Methotrexate and Metformin in Rheumatoid Arthritis Patients
Acronym: METorMET²
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry for Health and Solidarity, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2016/44
Record Dates: First submitted 2019-12-05; First posted 2019-12-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Arthritis, Rheumatoid
Keywords: rheumatoid arthritis; methotrexate; metformin; clinical trial
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Masking Description: placebo-controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental)
  Interventions: Drug: Metformin treatment; Drug: Methotrexate treatment
- Control arm (Placebo Comparator)
  Interventions: Other: Placebo; Drug: Methotrexate treatment

INTERVENTIONS:
Drug: Metformin treatment — 1500 mg once a day, per os, during six months
  Arms: Experimental arm
Other: Placebo — per os, during six months
  Arms: Control arm
Drug: Methotrexate treatment — per os

SUMMARY:
Methotrexate (MTX) is the anchor drug for patients with rheumatoid arthritis (RA). Despite its marked efficacy and acceptable side effect profile, about 1/3 of patients failed to reach RA remission. Metformin is the first-line therapy for type 2 diabetes. Its antioxidative and anti-inflammatory properties make it a good candidate for the treatment of inflammatory diseases such as rheumatoid arthritis.

DETAILED DESCRIPTION:
Methotrexate is usually the first-line disease modifying antirheumatic drugs (DMARD) for the treatment of RA. The main goal of its treatment is to reach disease remission but, despite its good efficacy, 1/3 of patients failed to achieve it. This could lead to the introduction of a biologic therapy which is more expensive and exposes the patient to a greater infection risk. Neutrophils through expulsion of neutrophil extracellular traps (NETs), were found to be important in RA pathogenesis (source of anti-citrullinated protein antibodies, activation of fibroblast-like synoviocytes…). The formation of NETs is reactive oxygen species (ROS) dependent, while metformin can selectivity inhibit mitochondrial respiratory chain complex I and decrease NADPH oxidase activity, thus leading to a decrease in ROS production.

Metformin is the first-line therapy for type 2 diabetes. Recently, a study presented its potential impact in the treatment of systemic lupus erythematosus according to its metabolic properties and the inhibition of NETosis.

The aim of this study is to compare the efficacy of Methotrexate/Metformin vs. Methotrexate alone on the decrease of RA activity in MTX-naive patients, after 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old,
* Patient affected by RA according to American College of Rheumatology (ACR) 2010 criteria
* DAS28-ESR > 3.2
* Methotrexate naïve patients, or without any methotrexate intake for more than six months.
* Men who accept to take active contraception during the study and during six months after the end of the Methotrexate treatment. Partner of patient will be informed of teratogenicity of MTX and will be advised to be on effective contraceptives for all the study duration.

OR

* Women with a negative test of β-human chorionic gonadotropin (HCG) who accept to take active contraception during the study and during six months after the end of the Methotrexate treatment
* Patients without any Metformin previous therapy.
* Being affiliated to a health insurance system
* Having signed an informed consent form (later than the day of inclusion and before any examination required by the research)

Exclusion Criteria:

* Patient who present contraindications to treatment with Methotrexate or Metformin
* Patient with type 1 or type 2 diabetes
* Patient with daily corticosteroid treatment at a dosage ≥ 15 mg/day within four weeks before the inclusion
* History of allergy or intolerance to biguanide
* Presence of anemia (hemoglobin < 80 g/l), neutropenia (neutrophils count < 1500 mm3), lymphopenia (lymphocytes count < 750 mm3), thrombopenia (platelets < 100 000/mm3) or bone marrow hypoplasia.
* Renal insufficiency with clearance < 50 ml/mn
* Decompensated heart failure
* Uncontrolled heart history
* Severe respiratory insufficiency
* Hepatic insufficiency, or bilirubin level upper than 5mg/dl (85,5 µmol/l), or aspartate transaminase (ASAT) / alanine aminotransferase (ALAT) more than twice the standard level.
* Acute or chronic infection, such as tuberculosis or HIV
* Critical ischemia of the lower limbs
* Recent stroke
* Patient with pleural effusion, or ascites
* Patient with stomatitis, mouth ulcers, or active gastrointestinal ulcer.
* Patient with alcohol intoxication
* B12 Vitamin deficiency
* Patient performing or planning to perform a long-fasting period
* Pregnant or breastfeeding women
* Patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change of level of RA activity according to Disease Activity score on 28 joints (DAS28-ESR) | At baseline (Day 0) and 6 months after baseline

SECONDARY OUTCOMES:
Proportion of patients who reach remission | At 6 months, 12 months and 24 months after baseline (Day 0)
Proportion of patients with low disease activity (DAS-ESR < 3,2) | At 6 months after baseline (Day 0)
Proportion of patients for which a biologic treatment is introduced | At 6 months, 12 months and 24 months after baseline (Day 0)
Mean dosage of Methotrexate in the two groups of randomization | At 6 months, 12 months and 24 months after baseline (Day 0)
Proportion of patients who present a serious adverse event within the two groups | At 6 months after baseline (Day 0)
Evolution of functional assessment according to Health Assessment Questionnaire (HAQ) within the two groups | At baseline (Day 0), 1 month, 3 months, 6 months, 12 months and 24 months after baseline
Mean value of weight in kilograms in each randomization group | At baseline (Day 0), 6 months and 24 months after baseline
Mean value of waist circumference in centimeters in each randomization group | At baseline (Day 0), 6 months and 24 months after baseline
Mean value of fasting glycemia in g/l in each randomization group | At baseline (Day 0), 6 months and 24 months after baseline
Mean value of hemoglobin A1c level (HbA1c) in percentage in each randomization group | At baseline (Day 0), 6 months and 24 months after baseline
Mean value of cholesterol levels and triglycerides levels in g/l in each randomization group | At baseline (Day 0), 6 months and 24 months after baseline
Mean value of insulinemia in µUI/ml in each randomization group | At baseline (Day 0), 6 months and 24 months after baseline
Mean value of bilirubin in mg/l in each randomization group | At baseline (Day 0), 6 months and 24 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christophe RICHEZ, Prof, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, MD, PhD, Study Chair — University Hospital, Bordeaux
Locations (12):
- France (12):
  - CH de la Côte Basque - service de rhumatologie, Bayonne
  - CHU de Bordeaux - service de rhumatologie, Bordeaux
  - CHU de Brest - service de rhumatologie, Brest
  - CH de Cahors - service de rhumatologie, Cahors
  - Clinique de l'Infirmerie protestante de Lyon - service de rhumatologie, Caluire-et-Cuire
  - CHD de Vendée - service de rhumatologie, La Roche-sur-Yon
  - CH du Mans - service de rhumatologie, Le Mans
  - CH de Libourne - service de rhumatologie, Libourne
  - CHU de Montpellier - service de rhumatologie, Montpellier
  - CHR Orléans la Source - service de rhumatologie, Orléans
  - CH de Pau - service de rhumatologie, Pau
  - CHU de Toulouse - service de rhumatolgie, Toulouse